CLINICAL TRIAL: NCT01274728
Title: Pilot Study on PAclitaxel-eluting Balloon in Primary PCI in Amsterdam. A Clinical Evaluation, to Study the Feasibility and Safety of a Paclitaxel-eluting Balloon in Primary Percutaneous Coronary Intervention for Acute ST-elevation Myocardial Infarction.
Brief Title: PAclitaxel-eluting Balloon in Primary PCI in Amsterdam; Pilot Study
Acronym: PAPPA-pilot
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Dr. R.J. van der Schaaf, Cardiology department OLVG
Other Study IDs: wo 09.070
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Primary percutaneous coronary intervention; Drug-eluting balloon; Bivalirudin
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biochemistry, haematology
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ST-elevated myocardial infarction: Those with a condition of chestpain (or equal complains) and ECG changes confirming STEMI.
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention with at least use of drug-eluting balloon and if necessary cross-over to bail-out stenting with BMS.

SUMMARY:
This clinical evaluation will study the feasibility and safety of a CE-marked paclitaxel-eluting balloon in primary PCI in patients with a STEMI. Drug eluting balloons provide the potential advantage of delivering a anti-proliferative drug, without the disadvantage of leaving a coronary stent, in STEMI patients treated with primary PCI.

DETAILED DESCRIPTION:
Multiple randomized clinical trials and pooled analyses have shown improved clinical outcomes of primary PCI when compared with fibrinolytic therapy. Primary PCI for STEMI results in greater patency of the infarct-related artery (IRA) and lower rates of death, re-infarction, and stroke when compared with fibrinolysis. The use of coronary stents has reduced the need for repeat revascularization in patients treated with primary PCI. However, in the setting of STEMI this reduction in target lesion revascularization (TLR) did not reduce re-infarction rates or both short term and long-term mortality rates. This was confirmed by a large meta-analysis by De Luca et al, using 13 randomized trials and involving 6922 patients. In studies evaluating DES versus BMS in STEMI mortality rates are similar in patients treated with BMS or DES. Although TLR rates are reduced with the use of DES, there have been concerns about long-term delay of arterial healing produced by both the Cypher DES and Taxus DES and the associated risk of late stent thrombosis. Anti-proliferative drugs in DES used to prevent neointimal hyperplasia also prevent the formation of an epithelial surface at the inner side of stents causing possible stent malapposition and potentionally late stent thrombosis. A new approach in treatment of STEMI is now available by the development of a drug eluting balloon. These DEB can be used with or without additional stent placement. Potential advantages compared to DES are a more homogeneous drug distribution, short lasting exposure and a higher local drug dose. Moreover, when no additional stent is needed, it might reduce the need for long term aggressive anti-platelet therapy in order to prevent acute, late or very late stent thrombosis. In short, DEB provides the potential advantage of delivering a anti-proliferative drug, without the disadvantage of leaving a coronary stent, in STEMI patients treated with primary PCI. The use of DEB is already tested for treatment of de novo coronary lesions and in-stent restenosis and has been shown to be a feasible and safe.In this clinical evaluation the use of the CE-marked Paclitaxel-eluting balloon with provisional stenting for STEMI will be evaluated on top of current highest standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction eligible for primary PCI:

  * 20 min of chest-pain and at least 1 mm ST-elevation in at least two contiguous leads, a new left bundle branch block or a true posterior myocardial infarction
  * reperfusion is expected to be feasible within 12 hours after onset of complaints
* Infarct related artery eligible for PPCI including stent implantation. Diameter of IRA ≥ 2.5 mm, ≤ 4 mm.
* Infarction is caused by a de novo lesion in a native coronary artery

Exclusion Criteria:

* Age < 18
* Reperfusion not feasible within 12 hours after onset of complaints
* Failed thrombolysis
* Infarct related artery unsuitable for PCI
* Sub-acute stent thrombosis
* STEMI caused by in-stent re-stenosis
* Infarct related vessel / target vessel SVG or LIMA
* Contraindication or resistance for bivalirudin, fondaparinux ,aspirin, clopidogrel and/or prasugrel.
* Participation in another clinical study, interfering with this protocol
* Cardiogenic shock prior to inclusion
* Uncertain neurological outcome e.g. resuscitation
* Intubation/ventilation
* Known intracranial disease (mass, aneurysm, AVM, hemorrhagic CVA, ischemic CVA/TIA < 6 months prior to inclusion or ischemic CVA with permanent neurological deficit)
* Gastro-intestinal / urinary tract bleeding < 2 months prior to inclusion
* Refusal to receive blood transfusion
* Platelet number < 100.000 x 10^9/L
* Planned major surgery within 6 weeks
* Stent implantation < 1 month prior to inclusion
* Expected mortality from any cause within the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are presented at the emergency room or in ambulance with STEMI
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-11

PRIMARY OUTCOMES:
Major acute coronary event | 1 month
  Defined as
  1. any death in which cardiac cause can not be excluded (death due to proximate cardiac cause, unwitnessed death, death of unknown cause, all procedure-related deaths)
  2. recurrent MI in the target vessel area (if no infarct localization is identified it is regarded target vessel related)
  3. target lesion revascularization (PCI within 5mm of the balloon(stent) area borders or CABG of the target vessel)

SECONDARY OUTCOMES:
Cross-over to bail-out stenting | 1, 6 and 12 months
Death from any cause | 1, 6 and 12 months
Major acute coronary event | 6 and 12 months
  Defined as
  1. any death in which cardiac cause can not be excluded (death due to proximate cardiac cause, unwitnessed death, death of unknown cause, all procedure-related deaths)
  2. recurrent MI in the target vessel area (if no infarct localization is identified it is regarded target vessel related)
  3. target lesion revascularization (PCI within 5mm of the balloon(stent) area borders or CABG of the target vessel)
In-hospital major acute coronary event | index hospitalisation
  Defined as, in-hospital index event:
  1. any death in which cardiac cause can not be excluded (death due to proximate cardiac cause, unwitnessed death, death of unknown cause, all procedure-related deaths)
  2. recurrent MI in the target vessel area (if no infarct localization is identified it is regarded target vessel related)
  3. target lesion revascularization (PCI within 5mm of the balloon(stent) area borders or CABG of the target vessel)
Recurrent MI non-target vessel related | 1, 6 and 12 months
Target vessel revascularisation | 1, 6 and 12 months
  Target vessel revascularisation, but not target lesion revasularisation (is primary outcome measure)
Stroke | 1, 6 and 12 months
  objectified and documented by a physician
Stent thrombosis | index hospitalisation, 1, 6 and 12 months
  according tot the ARC criteria
NON-CABG major bleeding | 1 month
  as in HORIZON trial
Hemorrhagic events | 1 month
  according to TIMI bleeding classification

CONTACTS AND LOCATIONS:
Overall Officials: R.J. van der Schaaf, MD, PhD, Principal Investigator — Onze Lieve Vrouwe Gasthuis Amsterdam; M.T. Dirksen, MD, PhD, Principal Investigator — Onze Lieve Vrouwe Gasthuis Amsterdam; N.S. Vos, MD, Study Chair — Onze Lieve Vrouwe Gasthuis Amsterdam; J.P.H. Herrman, MD, PhD, Study Director — Onze Lieve Vrouwe Gasthuis
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, Netherlands

REFERENCES:
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Zijlstra F, Hoorntje JC, de Boer MJ, Reiffers S, Miedema K, Ottervanger JP, van 't Hof AW, Suryapranata H. Long-term benefit of primary angioplasty as compared with thrombolytic therapy for acute myocardial infarction. N Engl J Med. 1999 Nov 4;341(19):1413-9. doi: 10.1056/NEJM199911043411901. PMID 10547403
- [Background] De Luca G, Suryapranata H, Stone GW, Antoniucci D, Biondi-Zoccai G, Kastrati A, Chiariello M, Marino P. Coronary stenting versus balloon angioplasty for acute myocardial infarction: a meta-regression analysis of randomized trials. Int J Cardiol. 2008 May 7;126(1):37-44. doi: 10.1016/j.ijcard.2007.03.112. Epub 2007 Jun 4. PMID 17544528
- [Background] Laarman GJ, Suttorp MJ, Dirksen MT, van Heerebeek L, Kiemeneij F, Slagboom T, van der Wieken LR, Tijssen JG, Rensing BJ, Patterson M. Paclitaxel-eluting versus uncoated stents in primary percutaneous coronary intervention. N Engl J Med. 2006 Sep 14;355(11):1105-13. doi: 10.1056/NEJMoa062598. PMID 16971717
- [Background] Spaulding C, Henry P, Teiger E, Beatt K, Bramucci E, Carrie D, Slama MS, Merkely B, Erglis A, Margheri M, Varenne O, Cebrian A, Stoll HP, Snead DB, Bode C; TYPHOON Investigators. Sirolimus-eluting versus uncoated stents in acute myocardial infarction. N Engl J Med. 2006 Sep 14;355(11):1093-104. doi: 10.1056/NEJMoa062006. PMID 16971716
- [Background] De Luca G, Stone GW, Suryapranata H, Laarman GJ, Menichelli M, Kaiser C, Valgimigli M, Di Lorenzo E, Dirksen MT, Spaulding C, Pittl U, Violini R, Percoco G, Marino P. Efficacy and safety of drug-eluting stents in ST-segment elevation myocardial infarction: a meta-analysis of randomized trials. Int J Cardiol. 2009 Apr 3;133(2):213-22. doi: 10.1016/j.ijcard.2007.12.040. Epub 2008 Apr 3. PMID 18394731
- [Background] Brar SS, Leon MB, Stone GW, Mehran R, Moses JW, Brar SK, Dangas G. Use of drug-eluting stents in acute myocardial infarction: a systematic review and meta-analysis. J Am Coll Cardiol. 2009 May 5;53(18):1677-89. doi: 10.1016/j.jacc.2009.03.013. PMID 19406344
- [Background] Degertekin M, Serruys PW, Tanabe K, Lee CH, Sousa JE, Colombo A, Morice MC, Ligthart JM, de Feyter PJ. Long-term follow-up of incomplete stent apposition in patients who received sirolimus-eluting stent for de novo coronary lesions: an intravascular ultrasound analysis. Circulation. 2003 Dec 2;108(22):2747-50. doi: 10.1161/01.CIR.0000103666.25660.77. Epub 2003 Nov 24. PMID 14638542
- [Background] McFadden EP, Stabile E, Regar E, Cheneau E, Ong AT, Kinnaird T, Suddath WO, Weissman NJ, Torguson R, Kent KM, Pichard AD, Satler LF, Waksman R, Serruys PW. Late thrombosis in drug-eluting coronary stents after discontinuation of antiplatelet therapy. Lancet. 2004 Oct 23-29;364(9444):1519-21. doi: 10.1016/S0140-6736(04)17275-9. PMID 15500897
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Two year follow-up after treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. Clin Res Cardiol. 2008 Oct;97(10):773-81. doi: 10.1007/s00392-008-0682-5. Epub 2008 Jun 5. PMID 18536865
- [Background] Unverdorben M, Vallbracht C, Cremers B, Heuer H, Hengstenberg C, Maikowski C, Werner GS, Antoni D, Kleber FX, Bocksch W, Leschke M, Ackermann H, Boxberger M, Speck U, Degenhardt R, Scheller B. Paclitaxel-coated balloon catheter versus paclitaxel-coated stent for the treatment of coronary in-stent restenosis. Circulation. 2009 Jun 16;119(23):2986-94. doi: 10.1161/CIRCULATIONAHA.108.839282. Epub 2009 Jun 1. PMID 19487593
- [Background] Unverdorben M, Kleber FX, Heuer H, Figulla HR, Vallbracht C, Leschke M, Cremers B, Hardt S, Buerke M, Ackermann H, Boxberger M, Degenhardt R, Scheller B. Treatment of small coronary arteries with a paclitaxel-coated balloon catheter. Clin Res Cardiol. 2010 Mar;99(3):165-74. doi: 10.1007/s00392-009-0101-6. Epub 2010 Jan 6. PMID 20052480
- [Background] Stone GW, Witzenbichler B, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Kornowski R, Hartmann F, Gersh BJ, Pocock SJ, Dangas G, Wong SC, Kirtane AJ, Parise H, Mehran R; HORIZONS-AMI Trial Investigators. Bivalirudin during primary PCI in acute myocardial infarction. N Engl J Med. 2008 May 22;358(21):2218-30. doi: 10.1056/NEJMoa0708191. PMID 18499566
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Vranckx P, Kint PP, Morel MA, Van Es GA, Serruys PW, Cutlip DE. Identifying stent thrombosis, a critical appraisal of the academic research consortium (ARC) consensus definitions: a lighthouse and as a toe in the water. EuroIntervention. 2008 Aug;4 Suppl C:C39-44. No abstract available. PMID 19202690